CLINICAL TRIAL: NCT03266289
Title: Evaluation of Short Term Outcome of Different Bifurcation Stenting Techniques at Assuit University Cath. Lab
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: MA Abdelreheem (Other)
Responsible Party: Sponsor-Investigator, MA Abdelreheem, Resident doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 17100301
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Unstable Angina
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary aim: evaluation of the short term outcome of different techniques used in bifurcational coronary arteries intervention regarding major adverse cardiac event (MACE): cardiac death, myocardial infarction, target vessel revascularization, or stent thrombosis and occurrence of Unstable angina (UA) with ECG changes and echo findings in the same target vessel in Assiut university Cath. lab.

Secondary aim: calculation of the percentage of bifurcational coronary arteries intervention in Assiut University Cath.lab

DETAILED DESCRIPTION:
IntroductionCoronary artery bifurcation lesions comprise one of the more complex lesion subsetsroutinely faced in interventional cardiology, accounting for up to 20% of all coronarydiseases treated by percutaneous coronary intervention (PCI) The technical difficulties inherent in the treatment of bifurcation lesions, associatedwith their lower success and higher complication rates compared with non-bifurcationlesions, have always been the object of intense research activity, with publication ofcontemporary studies in the past few years contributing significantly to the decisionmaking process.Bifurcation lesions are challenging to categorize, since they are variable not only intheir anatomy (location of plaque, plaque burden, angle between branches, site ofbifurcation, and size of branches), but also in the dynamic anatomic changes duringtreatment caused by dissections and carina shift. Despite these challenges complicatingclassification of bifurcation lesions, many definitions have been proposed in an effort tounify this common clinical situation. A coronary bifurcation lesion is defined as (coronary artery narrowing occurringadjacent to, and/or involving, the origin of a significant side branch). A significant sidebranch (SB) is a branch that, if lost, can impact the prognosis of the patient. General different classifications of coronary bifurcation lesions have been proposed, dueto the variety of possible bifurcation lesions, with different technical implications,treatment options, and prognosis. The most used, for its simplicity and reproducibility,is the Medina classification. This classification is based on the presence or absence ofnarrowing >50% on each of the three components of the bifurcation: the main branchproximal (MBP), the main branch distal, and the SB. A value of 0 or 1 is assigned toeach of the three segments in the following order: MBP, main branch distal, and SB. Forexample, a bifurcation lesion involving the MBP and the SB would be defined as 1, 0,1. Seven morphologies are therefore possible. Despite being the most usedclassification, the Medina has several limitations, since it does not consider the plaqueburden, branch diameter, lesion length, bifurcation angles, the presence of ostialdisease, or calcification.

The goal of percutaneous coronary intervention in bifurcation lesions is tomaximize flow in the main branch (MB), maintain flow in the SB, prevent its occlusion,and maximize long-term patency. Data about bifurcational lesions percentage and short term outcome of differenttechniques used in intervention in our cath lab is still unknown.Aim of the study

ELIGIBILITY:
Inclusion Criteria:

* All patients with true bifurcational coronary arteries lesion defined as (lesions in which there is more than 50% diameter stenosis in both the parent vessel and the ostium of the side branch arising from the lesion, and both are more than 2.0 mm in diameter by visual estimation) (13) undergoing intervention either urgent or elective in Assiut university Cath. lab during period from September 2017 to September 2018 will be included in this study.

Exclusion Criteria:

* • Contraindications to PCI of bifurcation lesions would be any patient unwilling to undergo PCI, coronary anatomy that is not amenable to PCI (e.g., small caliber with diffuse disease), intermediate lesions in the absence of symptoms, and/or subjective evidence of ischemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include patients diagnosed as bifurcational coronary arteries Iesion underwent intervention
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary aim: evaluation of the short term outcome of different techniques used in bifurcational coronary arteries intervention | 1 year
  Primary aim: evaluation of the short term outcome of different techniques used in bifurcational coronary arteries intervention regarding major adverse cardiac event (MACE): cardiac death, myocardial infarction, target vessel revascularization, or stent

SECONDARY OUTCOMES:
Secondary aim: calculation of the percentage of bifurcational coronary arteries intervention in Assiut University Cath.lab | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amr A. Youssef, Prof doctor, Study Director — Assiut University; Mohamed A. Abdelhafez, Doctor, Study Director — Assiut University